CLINICAL TRIAL: NCT05653895
Title: Independent and Additive Effects Of Micronutrients With Metformin In Patients With PCOS:A Double Blind Randomized Placebo Controlled Trial
Brief Title: Independent and Additive Effects Of Micronutrients With Metformin In Patients With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Medical University Peshawar (Other)
Responsible Party: Principal Investigator, Mohsin Shah, Assistant Professor, Khyber Medical University Peshawar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KhyberMU
Record Dates: First submitted 2022-03-01; First posted 2022-12-16 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: PCOS
MeSH Terms: interventions — Resveratrol; Metformin; Arginine; Ubiquinone

STUDY DESIGN:
Intervention Model Description: Treatment of PCOS with Metformin vs Combination therapy
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Triple (Participant ,Care provider ,Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Active Comparator): Resveratrol (2 gm daily) 50 patients with PCOS will receive Resveratrol 1000mg BD daily
  Interventions: Dietary Supplement: Resveratrol
- Arm 2 (Active Comparator): Metformin (1000mg daily),Resveratrol(2 gm daily) 50 patients with PCOS will receive Metformin 500mg,Resveratrol 1000 mg BD daily
  Interventions: Dietary Supplement: Resveratrol; Drug: Metformin
- Arm 3 (Active Comparator): L-Arginine(3 gm daily), Acetyl L-Carnitine (3 gm daily),CoQ10(200 mg daily) 50 patients with PCOS will receive L Arginine 1500mg,Acetyl L Carnitine 1500mg ,COQ10 100mg BD daily respectively
  Interventions: Combination Product: Acetyl-L-Carnitin, L Arginine, Co-Q10
- Arm 4 (Active Comparator): L-Arginine(3 gm daily), Acetyl L-Carnitine (3 gm daily),CoQ10(200 mg daily),Metformin (1000mg daily) 50 patients with PCOS will receive L Arginine 1500mg,Acetyl L Carnitine 1500mg,COQ10 100mg BD daily respectively
  Interventions: Drug: Metformin; Combination Product: Acetyl-L-Carnitin, L Arginine, Co-Q10

INTERVENTIONS:
Dietary Supplement: Resveratrol — Resveratrol
  Arms: Arm 1; Arm 2
Drug: Metformin — Metformin
  Arms: Arm 2; Arm 4
Combination Product: Acetyl-L-Carnitin, L Arginine, Co-Q10 — Treatment of PCOS with combination of Acetyl-L-Carnitin, L Arginine, Co-Q10
  Arms: Arm 3; Arm 4

SUMMARY:
The investigators aim to conduct a double blind randomized clinical trial to study the independent and additive effects of micronutrients (Resveratrol, Acetyl-L Carnitine, L Arginine and COQ10 ) with Metformin in patients with PCOS .Women diagnosed with PCOS according to National Institute of Health( NIH) 2012 extension of European Society of Human Reproduction and Embryology /American Society of Reproductive Medicine ESHRE /ASRM 2003 criteria will be included according to a specific phenotype including Hyperandrogenism, Ovulatory dysfunction and Polycystic Ovarian Morphology. The investigators propose that by using combination therapy with micro supplements like Resveratrol, Acetyl-L Carnitine, L Arginine and COQ10 will produce greater improvement better than or at least comparable to Metformin in metabolic and endocrine profile of patients with PCOS.

DETAILED DESCRIPTION:
Polycystic ovary syndrome is a condition which is manifested by certain polycystic ovarian morphologic features, hyperandrogenism and ovulatory dysfunction. As per the revised diagnostic criteria by National Institute of Health 2012, about 6 to 10% women of the reproductive age are affected by the classic polycystic ovarian syndrome, the prevalence of which is twice as more according to the broader Rotterdam standards . One important cause of distress in patients with this syndrome is the excessive expression of androgens (e.g., hirsutism) which leads to infertility. A number of reports based on PCOS suggest that genetic anomalies of follicular maturation and ovarian steroidogenesis also have a crucial role in the development and occurrence of PCOS. This disorder is polygenic in nature and contributes towards metabolic diseases like obesity . About 50 to 80% women having PCOS are obese . Not only has this but PCOS also had a connection with an elevated risk of cardiovascular disease . Type-2 diabetes amongst women with this syndrome is reported to be 8 to 10%, and the compromised glucose tolerance cases are reported as high as 30 to 35% of US. Moreover, the chances of occurrence of this disease is highly associated with changes in age, history of diabetes in family and obesity . PCOS is a multifaceted health issue having several short and long term effects on woman's health. These include cardiovascular diseases, metabolic and sexual dysfunction, depression and anxiety that effects the overall quality of life. The present study documents the impact of PCOS and its complications on overall quality of life and how new treatment options can help minimize the signs and symptoms associated with the disease condition. Some of the recent focused therapeutic compounds reported in this context are Resveratrol, L-Carnitine, Co-Q10, L-Arginine and Decanoic acid as naturally occurring nutraceuticals and metformin as standard therapeutic drug against PCOS.

Resveratrol (3,5,4-trihydroxystilbene)-A naturally occurring polyphenol, found in grapes, peanuts, red wine and many medicinal plants . According to studies, this compound may have many antidiabetic, anti-inflammatory and antioxidant actions . Kong et al. highlighted that resveratrol decreases the atretic follicles which significantly increase the number of oocytes . This leads to an inhibition of both, apoptosis and primordial to the developing follicle in rats of different age groups . Resveratrol has been reported to interact with multiple cell targets, but its major effects are brought about by the activation of SIRT1 (silent information regulator 1) . SIRT1, which is a key player in energy metabolism and homeostasis, is a mammalian homologue of Sir2 (yeast) which deacetylates many mammalian cell targets. The SIRT1 is basically expressed in oocytes and human granulosa nuclei cells at multiple developmental stages of the follicles. It is also responsible for suppressing inflammation. Moreover, SIRT1 is also involved in protecting the oocytes from age dependent insufficiencies through oxidative stress . Resveratrol has a tendency to suppress inflammation by activating SIRT1 and as a result the symptoms of inflammation are reduced in many autoimmune disease models like rheumatoid arthritis, colitis, encephalomyelitis and type I diabetes L-Carnitine is involved in fatty acid oxidation by long chain fatty acids transport inside the mitochondria for oxidation to produce metabolic energy and have effects on glucose metabolism in tissues. L-Carnitine is known to regulate energy production . Studies have shown that patients treated with L-Carnitine have improved ovulation and pregnancy rates and is very well tolerated by the patients .

Coenzyme Q10 (CoQ10) a lipid soluble coenzyme which is an important component of the inner membrane of mitochondria. It is a key regulator of oxidative phosphorylation in the electron transport chain for ATP synthesis. A number of studies have reported a protective role of CoQ10 in ovaries by restoring aging of ovaries and improving mitochondrial function . According to a recent finding, administration of 20 mg/kg of CoQ10 in a rat model led to increased insulin sensitivity, suggesting its antidiabetic potential .

Decanoic acid- is naturally occurring fatty acid present in palm and coconut oils . Lee et al suggested that decanoic acid along with metformin altered cAMP signaling and normalized the androgen synthesis. Moreover, in a diabetic mouse model, treatment with decanoic acid led to improved glucose sensitivity. In another study, letrozole-induced rat PCOS model, the administration of decanoic acid reduced the levels of androgen and 3-HSD which led to restoration of the estrous cycle . These studies suggest a positive role of decanoic acid in management and treatment of insulin resistance and hyperandrogenism in PCOS patients.

L-Arginine is an amino acid that plays a role in a number of metabolic pathways and serves as a substrate for NOS (Nitric Oxide synthase) enzyme which is essentially involved in normal insulin signaling and endothelial function . In other findings, it is proposed that L-Arginine also enhances metabolic profile, β-cell function and has anti-oxidant potential . The ovarian health was also improved along with follicular growth, luteal function and oocyte development by the administration of L-Arginine. According to a previous study, PCOS patients had lowered levels of NO (nitric oxide) due to reduced expression of NOS which consequently led to a decline in arginine bioavailability. Therefore, L-arginine supplementation can have a therapeutic potential .

Metformin a biguanide which is used in type 2 diabetes and is mostly used as a gold standard drug for PCOS therapy . The mechanism of action is such that it helps in inhibition of hepatic gluconeogenesis and intestinal glucose absorption which ultimately improves insulin signaling .

Metformin has a direct and important role in human ovarian steroidogenesis. It inhibits insulin stimulated progesterone and gonadotrophin dose dependently in granulosa cells . According to a recent research report, it was reported that metformin treatment in infertile, anovulatory PCOS women, resulted in pregnancy, higher ovulation and live birth rates as compared to placebo . PCOS is a systemic condition, an endocrinopathy whose etiology is still not understood, correct treatment regimens of PCOS will not only improve menstrual cycle irregularities of the patients but will also improve the metabolic or endocrinological parameters . PCOS sufferers are also known to have increased levels of perceived stress which will be considered in the study. Very little evidence is available on combination therapy for treatment of PCOS patients. In this study the investigators goal will be to come up with a better treatment option to treat the disease effectively.

ELIGIBILITY:
Inclusion Criteria:

* PCOS women aged 16 -45 years.Diagnosis of PCOS will be made according to NIH 2012 extension of ESHRE/ASRM 2003 criteria Identification of specific phenotype will be included

  1. HA+OD+PCOM (Hyperandrogenism, Ovulatory dysfunctions, Polycystic ovarian morphology)
  2. HA+OD
  3. HA+PCOM
  4. PCOM+OD

Exclusion Criteria:

1. Women with hyperprolactenemia
2. Diabetes Mellitus
3. Cushing syndrome
4. Androgen secreting tumours
5. Non classical congenital adrenal hyperplasia
6. History of seizures
7. Patients on anti coagulants, anti platelets ,isoproterenol ,antidepressants, potassium sparing diuretics
8. Pregnancy or use of contraceptives
9. Patients with thyroid disease
10. Patients on hormonal therapy -

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-02-07 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 6 months
  PCOS associated insulin resistance and hyperinsulinemia by HOMA-IR
Menstural Irregularities | 6 months
  Oligo/Anovulation, Questionnaire based history taking of each participant
Anti mullerian Hormone | 6 months
  Measurement of Anti mullerian hormone by ELISA
Dehydroepiandrosterone | 6 months
  Measurement of Dehydroepiandrosterone using ELISA

SECONDARY OUTCOMES:
Antioxidant Assays | 6 months
  Measuring Total AntiOxidant Capacity by FRAP ASSAY
Anti oxidant Assays | 6 months
  Measuring MDA (Malondialdehyde) by TBARS
Mental health questionnaire | 6 months
  Will be assessed by using Polycystic Ovarian Syndrome Quality Of Life Tool
Molecular characterisation | 6 months
  SNP genotyping of THADA and DENNDIA
perceived stress response (PSS-14) questionnaire | 6 months
  Stress response
profile of mood stress (POMS) by structured questionnaire | 6 months
  Stress response

CONTACTS AND LOCATIONS:
Overall Officials: Mohsin Shah, PHD, Principal Investigator — Department of Physiology ,Khyber Medical University ,Peshawar, Pakistan
Locations (1):
- Bacha Khan Medical Complex Swabi, Swabi, Khyber Pukhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dumesic DA, Oberfield SE, Stener-Victorin E, Marshall JC, Laven JS, Legro RS. Scientific Statement on the Diagnostic Criteria, Epidemiology, Pathophysiology, and Molecular Genetics of Polycystic Ovary Syndrome. Endocr Rev. 2015 Oct;36(5):487-525. doi: 10.1210/er.2015-1018. PMID 26426951
- [Background] Wild RA, Carmina E, Diamanti-Kandarakis E, Dokras A, Escobar-Morreale HF, Futterweit W, Lobo R, Norman RJ, Talbott E, Dumesic DA. Assessment of cardiovascular risk and prevention of cardiovascular disease in women with the polycystic ovary syndrome: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society. J Clin Endocrinol Metab. 2010 May;95(5):2038-49. doi: 10.1210/jc.2009-2724. Epub 2010 Apr 7. PMID 20375205
- [Background] Ehrmann DA, Barnes RB, Rosenfield RL, Cavaghan MK, Imperial J. Prevalence of impaired glucose tolerance and diabetes in women with polycystic ovary syndrome. Diabetes Care. 1999 Jan;22(1):141-6. doi: 10.2337/diacare.22.1.141. PMID 10333916
- [Background] Legro RS, Kunselman AR, Dodson WC, Dunaif A. Prevalence and predictors of risk for type 2 diabetes mellitus and impaired glucose tolerance in polycystic ovary syndrome: a prospective, controlled study in 254 affected women. J Clin Endocrinol Metab. 1999 Jan;84(1):165-9. doi: 10.1210/jcem.84.1.5393. PMID 9920077
- [Background] Ortega I, Duleba AJ. Ovarian actions of resveratrol. Ann N Y Acad Sci. 2015 Aug;1348(1):86-96. doi: 10.1111/nyas.12875. PMID 26315293
- [Background] Rege SD, Kumar S, Wilson DN, Tamura L, Geetha T, Mathews ST, Huggins KW, Broderick TL, Babu JR. Resveratrol protects the brain of obese mice from oxidative damage. Oxid Med Cell Longev. 2013;2013:419092. doi: 10.1155/2013/419092. Epub 2013 Sep 15. PMID 24163719
- [Background] Guo S, Yao Q, Ke Z, Chen H, Wu J, Liu C. Resveratrol attenuates high glucose-induced oxidative stress and cardiomyocyte apoptosis through AMPK. Mol Cell Endocrinol. 2015 Sep 5;412:85-94. doi: 10.1016/j.mce.2015.05.034. Epub 2015 Jun 6. PMID 26054749
- [Background] Kong XX, Fu YC, Xu JJ, Zhuang XL, Chen ZG, Luo LL. Resveratrol, an effective regulator of ovarian development and oocyte apoptosis. J Endocrinol Invest. 2011 Dec;34(11):e374-81. doi: 10.3275/7853. Epub 2011 Jul 7. PMID 21738004
- [Background] Borra MT, Smith BC, Denu JM. Mechanism of human SIRT1 activation by resveratrol. J Biol Chem. 2005 Apr 29;280(17):17187-95. doi: 10.1074/jbc.M501250200. Epub 2005 Mar 4. PMID 15749705
- [Background] Lee D, Goldberg AL. SIRT1 protein, by blocking the activities of transcription factors FoxO1 and FoxO3, inhibits muscle atrophy and promotes muscle growth. J Biol Chem. 2013 Oct 18;288(42):30515-30526. doi: 10.1074/jbc.M113.489716. Epub 2013 Sep 3. PMID 24003218
- [Background] Xuzhu G, Komai-Koma M, Leung BP, Howe HS, McSharry C, McInnes IB, Xu D. Resveratrol modulates murine collagen-induced arthritis by inhibiting Th17 and B-cell function. Ann Rheum Dis. 2012 Jan;71(1):129-35. doi: 10.1136/ard.2011.149831. Epub 2011 Sep 27. PMID 21953348
- [Background] Bentinger M, Brismar K, Dallner G. The antioxidant role of coenzyme Q. Mitochondrion. 2007 Jun;7 Suppl:S41-50. doi: 10.1016/j.mito.2007.02.006. Epub 2007 Mar 16. PMID 17482888
- [Background] Amin MM, Asaad GF, Abdel Salam RM, El-Abhar HS, Arbid MS. Novel CoQ10 antidiabetic mechanisms underlie its positive effect: modulation of insulin and adiponectine receptors, Tyrosine kinase, PI3K, glucose transporters, sRAGE and visfatin in insulin resistant/diabetic rats. PLoS One. 2014 Feb 20;9(2):e89169. doi: 10.1371/journal.pone.0089169. eCollection 2014. PMID 24586567
- [Background] Elson CE. Tropical oils: nutritional and scientific issues. Crit Rev Food Sci Nutr. 1992;31(1-2):79-102. doi: 10.1080/10408399209527562. PMID 1345319
- [Background] Malapaka RRV, Khoo S, Zhang J, Choi JH, Zhou XE, Xu Y, Gong Y, Li J, Yong EL, Chalmers MJ, Chang L, Resau JH, Griffin PR, Chen YE, Xu HE. Identification and mechanism of 10-carbon fatty acid as modulating ligand of peroxisome proliferator-activated receptors. J Biol Chem. 2012 Jan 2;287(1):183-195. doi: 10.1074/jbc.M111.294785. Epub 2011 Oct 28. PMID 22039047
- [Background] Wu G, Bazer FW, Davis TA, Kim SW, Li P, Marc Rhoads J, Carey Satterfield M, Smith SB, Spencer TE, Yin Y. Arginine metabolism and nutrition in growth, health and disease. Amino Acids. 2009 May;37(1):153-68. doi: 10.1007/s00726-008-0210-y. Epub 2008 Nov 23. PMID 19030957
- [Background] Boger RH. The pharmacodynamics of L-arginine. J Nutr. 2007 Jun;137(6 Suppl 2):1650S-1655S. doi: 10.1093/jn/137.6.1650S. PMID 17513442
- [Background] Piatti PM, Monti LD, Valsecchi G, Magni F, Setola E, Marchesi F, Galli-Kienle M, Pozza G, Alberti KG. Long-term oral L-arginine administration improves peripheral and hepatic insulin sensitivity in type 2 diabetic patients. Diabetes Care. 2001 May;24(5):875-80. doi: 10.2337/diacare.24.5.875. PMID 11347747
- [Background] Victor VM, Rocha M, Banuls C, Alvarez A, de Pablo C, Sanchez-Serrano M, Gomez M, Hernandez-Mijares A. Induction of oxidative stress and human leukocyte/endothelial cell interactions in polycystic ovary syndrome patients with insulin resistance. J Clin Endocrinol Metab. 2011 Oct;96(10):3115-22. doi: 10.1210/jc.2011-0651. Epub 2011 Jul 21. PMID 21778215
- [Background] Velazquez EM, Mendoza S, Hamer T, Sosa F, Glueck CJ. Metformin therapy in polycystic ovary syndrome reduces hyperinsulinemia, insulin resistance, hyperandrogenemia, and systolic blood pressure, while facilitating normal menses and pregnancy. Metabolism. 1994 May;43(5):647-54. doi: 10.1016/0026-0495(94)90209-7. PMID 8177055
- [Background] An H, He L. Current understanding of metformin effect on the control of hyperglycemia in diabetes. J Endocrinol. 2016 Mar;228(3):R97-106. doi: 10.1530/JOE-15-0447. Epub 2016 Jan 7. PMID 26743209
- [Background] Mansfield R, Galea R, Brincat M, Hole D, Mason H. Metformin has direct effects on human ovarian steroidogenesis. Fertil Steril. 2003 Apr;79(4):956-62. doi: 10.1016/s0015-0282(02)04925-7. PMID 12749437
- [Background] Morley LC, Tang T, Yasmin E, Norman RJ, Balen AH. Insulin-sensitising drugs (metformin, rosiglitazone, pioglitazone, D-chiro-inositol) for women with polycystic ovary syndrome, oligo amenorrhoea and subfertility. Cochrane Database Syst Rev. 2017 Nov 29;11(11):CD003053. doi: 10.1002/14651858.CD003053.pub6. PMID 29183107
- [Derived] Zahra M, Shah M, Iqbal F, Zubair T, Habib R, Zulfiqar F. Efficacy Of Combined Nutritional And Pharmacological Interventions In PCOS: A Six Month Randomized Controlled Trial. Naunyn Schmiedebergs Arch Pharmacol. 2025 Sep 30. doi: 10.1007/s00210-025-04626-6. Online ahead of print. PMID 41026176